CLINICAL TRIAL: NCT07310628
Title: Comparison of Analgesic Efficacy of Intrathecal Levobupivacaine With and Without Oral Tizanidine in Lower Limb Surgeries: A Prospective Randomized Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: All India Institute of Medical Sciences, Raebareli, UP (Unknown)
Responsible Party: Principal Investigator, ADABALA VIJAY BABU, ABabu, All India Institute of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 15
Record Dates: First submitted 2025-11-19; First posted 2025-12-30 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Tizanididne; Levobupicaine; Lower Limb Surgery; Pain, Chronic
Keywords: tizanidine
MeSH Terms: conditions — Chronic Pain | interventions — tizanidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tizanidine group (Experimental): Group T received 3 ml of 0.5% hyperbaric levobupivacaine and 4 mg of oral tizanidine 1 hour before surgery
  Interventions: Drug: Tizanidine
- placebo (Placebo Comparator): No active drug will be given per oral
  Interventions: Drug: Tizanidine

INTERVENTIONS:
Drug: Tizanidine — Group T received 3 ml of 0.5% hyperbaric levobupivacaine and 4 mg of oral tizanidine 1 hour before surgery

SUMMARY:
Tizanidine, alpha-2 adrenergic receptor agonist, provides analgesic and hemodynamic benefits, which could enhance the efficacy of local anaesthetics. This randomized controlled trial examines the effectiveness of oral tizanidine as an adjunct to intrathecal levobupivacaine for spinal anaesthesia in lower limb surgeries

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 to 60 years with an ASA grade of I-II, who were scheduled for elective lower limb surgeries with a duration of less than 2 hours and 30 mins.

Exclusion Criteria:

* Patients with certain conditions such as pregnancy, coagulopathy, cerebrovascular disease, systemic infections, inability to understand the study protocol, allergy to local anaesthetics, psychiatric disorders affecting evaluation, infection at the injection site, kidney and liver diseases, myelopathy or peripheral neuropathy, spinal stenosis, prior spinal surgeries, raised intracranial pressure, multiple sclerosis, spina bifida, those receiving thromboprophylaxis and refusal to participate in the study were excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-08-20 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Onset of action | intraoperative period after the spinal anaesthesia was given
  The duration of the sensory block was measured using the two-segment regression method, while the time until the first need for pain relief after surgery was used to determine the duration of analgesia. The modified Bromage scale was used to assess motor block. (0 = Ability to flex hips, knees, and ankles without paralysis; 1 = the ability to move the knees but not extend the legs; 2 = ability to flex at the ankles but not the knees; 3 = unable to move any part of the lower limb). The time between the injection and the highest Bromage score was used to determine the onset time of motor block.

SECONDARY OUTCOMES:
pain score | intraoperative and post operative period up to 24 hours
  Intraoperatively patients' Visual Analog Scale (VAS) scores were assessed. Post operatively VAS score will be assessed in PACU every 4th hourly up to 24 hours . The time to the first analgesic requirement was recorded, with tramadol (100 mg) administered when VAS scores exceeded 4. VAS score 0 is no pain and 10 is intense pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Adabala Vijay Babu, Raebareli, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Yes
if needed the data needed will be shared